CLINICAL TRIAL: NCT05417191
Title: Effect of Fish Consumption Enriched With Biologically Active Lipids From Olive Pomace, on Cardiovascular Risk Factors in Apparently Healthy Volunteers
Brief Title: Effect of Differently Fed Farmed Gilthead Sea Bream Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: Nireus Aquaculture (Unknown); National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Smaragdi Antonopoulou, Professor in Biochemistry, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25/07/2012
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cardiometabolic Health
Keywords: fish; sea bream; dietary intervention; olive oil; platelet aggregation; thrombosis; inflammation; cardioprotection
MeSH Terms: conditions — Thrombosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional fish (Active Comparator): This arm will consume 2 portions of gilthead seabream fed with conventional diet. Each portion weighed on average 380 g (raw, quantity of edible fillet approximately 170 g). Participants were instructed to consume fish twice weekly, one portion at a time.
  Interventions: Behavioral: Conventional fish
- Enriched fish (Experimental): This arm will consume 2 portions of gilthead seabream fed with olive pomace enriched diet. Each portion weighed on average 380 g (raw, quantity of edible fillet approximately 170 g). Participants were instructed to consume fish twice weekly, one portion at a time.
  Interventions: Behavioral: Enriched fish

INTERVENTIONS:
Behavioral: Conventional fish — Participants initially randomized to this intervention arm will be provided with conventional sea bream fillets and will be asked to consume them twice weekly for 8 weeks. Conventional sea bream fillets will be produced by a fish farming company using standard procedures. Participants will also be instructed to keep the reception of prescribed medications and dietary supplements stable and not to change their lifestyle habits (e.g. other dietary habits besides fish consumption, physical activity habits or sleep habits) during the intervention. After a 6-week wash-out period (no fish consumption), participants will cross over to the other intervention arm.
  Arms: Conventional fish
Behavioral: Enriched fish — Participants initially randomized to this intervention arm will be provided with conventional sea bream fillets and will be asked to consume them twice weekly for 8 weeks. Conventional sea bream fillets will be produced by a fish farming company using a diet enriched with olive pomace. Participants will also be instructed to keep the reception of prescribed medications and dietary supplements stable and not to change their lifestyle habits (e.g. other dietary habits besides fish consumption, physical activity habits or sleep habits) during the intervention. After a 6-week wash-out period (no fish consumption), participants will cross over to the other intervention arm.
  Arms: Enriched fish

SUMMARY:
The trial was a double-blind randomized dietary intervention study with a 1:1 allocation ratio, conducted in accordance with the Declaration of Helsinki. This study compared two treatments, i.e., farmed fish fed with olive pomace enriched diet (enriched fish; EF) versus farmed fish fed with fish oil diet (conventional fish; CF), using a crossover design. The study lasted 22 weeks; treatment period one (8 weeks, mid-January-end of March), washout period (6 weeks), and treatment period two (8 weeks, mid-May-end of July). The participants were equally distributed to the two treatments along treatment periods. Eligible subjects were all adults aged between 30 and 65 years old with a body mass index (BMI) between 24.0 and 31.0 kg/m2 who met the eligibility criteria for habitual fish consumption (<150 g of cooked fish per week). Exclusion criteria were pregnancy, current or recent weight loss effort, use of dietary supplements and being under treatment for any medical disorder. Subjects were allowed to use medical treatment for thyroid gland disorders, iron or folic acid supplements, contraceptives or hormone replacement therapy (HRT) for women, provided they would continue receiving their medication throughout the study. The aim of the study was to evaluate the effects of consumption of fillets from differently fed farmed gilthead sea bream on markers of cardiometabolic health such as platelet aggregation, circulating haemostatic markers, markers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 years old
* Body Mass Index between 24-31 kg/m^2
* Habitual fish consumption: <150 g of cooked fish per week

Exclusion Criteria:

* Pregnancy
* Current or recent weight loss effort
* Use of dietary supplements
* Being under treatment for any medical disorder

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline of adenosine diphosphate-induced platelet aggregation at 8 weeks | 0 (baseline) and 8 weeks
  Efficiency concentration fifty of adenosine diphosphate-induced platelet aggregation (microM) will be assessed by light transmittance aggregometry
Change from baseline of platelet activating factor-induced platelet aggregation at 8 weeks | 0 (baseline) and 8 weeks
  Efficiency concentration fifty of platelet activating factor-induced platelet aggregation (microM) will be assessed by light transmittance aggregometry
Change from baseline of thrombin-induced platelet aggregation at 8 weeks | 0 (baseline) and 8 weeks
  Efficiency concentration fifty of thrombin-induced platelet aggregation (microM) will be assessed by light transmittance aggregometry
Change from baseline in of plasminogen activator inhibitor-1 activity at 8 weeks | 0 (baseline) and 8 weeks
  Plasminogen activator inhibitor-1 activity (mAU/mL) will be measured in blood samples using commercially available ELISA kits
Change from baseline in soluble P-selectin levels at 8 weeks | 0 (baseline) and 8 weeks
  Soluble P-selectin levels (ng/mL) will be measured in blood samples using commercially available ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: Smaragdi Antonopoulou, PhD, Principal Investigator — Department of Nutrition and Dietetics, Harokopio University; Elizabeth Fragopoulou, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University; Tzortzis Nomikos, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University; Meropi D Kontogianni, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University; Michael Georgoulis, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University
Locations (1):
- Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared to investigators for the purpose of individual participant data meta-analysis, provided that the proposed use of the data has been approved by the Study Principal Investigator. Proposals should be directed to antonop@hua.gr. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Ntzouvani A, Antonopoulou S, Fragopoulou E, Kontogianni MD, Nomikos T, Mikellidi A, Xanthopoulou Mu, Kalogeropoulos N, Panagiotakos D. Effect of Differently Fed Farmed Gilthead Sea Bream Consumption on Platelet Aggregation and Circulating Haemostatic Markers among Apparently Healthy Adults: A Double-Blind Randomized Crossover Trial. Nutrients. 2021 Jan 20;13(2):286. doi: 10.3390/nu13020286. PMID 33498445